CLINICAL TRIAL: NCT03208842
Title: Relation of Implantation Site to Placental Site in Presence or Absence of Cesarean Section Scar With Doppler Assessment of Retro Chorionic Blood Flow
Brief Title: Relation of Implantation Site to Placental Site in Presence or Absence of Cesarean Section Scar
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Professor, Cairo University
Other Study IDs: 6
Record Dates: First submitted 2017-06-30; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Placenta Previa
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women with previous cesarean scar: the patient will be examined son graphically at 3 visits
  1. The first visit at less than 10 weeks gestation :trans vaginal ultrasound with partially filled bladder to nullify effect of anteversion of the uterus for assessment of
     ---the site of the intrauterine gestational sac in relation to the endometrial cavity .
     -----doppler assessment of the retro chorionic blood flow in the area behind the maximum chorionic tissue to detect sensitivity index (RI),in cases of low gestational sac Doppler assessment of peri trophoplastic blood flow will be assessed.
  2. then the patient will be enrolled during routine ANC till delivery and data collected at32-34 weeks gestation regarding placental site will be correlated with 1st data and data at delivery .
  Interventions: Radiation: trans vaginal ultrasound
- women without previous cesarean scar: the patient will be examined son graphically at 3 visits
  1. The first visit at less than 10 weeks gestation :trans vaginal ultrasound with partially filled bladder to nullify effect of anteversion of the uterus for assessment of
     ---the site of the intrauterine gestational sac in relation to the endometrial cavity .
     -----doppler assessment of the retro chorionic blood flow in the area behind the maximum chorionic tissue to detect sensitivity index (RI),in cases of low gestational sac Doppler assessment of peri trophoplastic blood flow will be assessed.
  2. then the patient will be enrolled during routine ANC till delivery and data collected at32-34 weeks gestation regarding placental site will be correlated with 1st data and data at delivery .
  Interventions: Radiation: trans vaginal ultrasound

INTERVENTIONS:
Radiation: trans vaginal ultrasound — trans vaginal ultrasound with partially filled bladder to nullify effect of anteversion of the uterus for assessment of
  ---the site of the intrauterine gestational sac in relation to the endometrial cavity

SUMMARY:
After gaining verbal consent , Patients included in this study will be subjected to:

1. history taking :

   * peronal history .
   * obstetric history.
   * past history
2. general examination including vital signs
3. abominal and pelvic examination
4. the patient will be examined son graphically at 3 visits

   1. The first visit at less than 10 weeks gestation :trans vaginal ultrasound with partially filled bladder to nullify effect of anteversion of the uterus for assessment of---the site of the intrauterine gestational sac in relation to the endometrial cavity . For the purposes of this study and to obtain consistent findings, it was decided to have only five subgroups of gestational site implantation in relation to the endometrial cavity (Fig. 2):

      1. anterior,
      2. posterior,
      3. Fundal,
      4. low-lying anterior,\
      5. low lying posterior We adopted the definition of implantation site from previous publication (Abdallah et al., 2012). The implantation site is visualized in the sagittal plane as a hyperechoic ring that occupies one side of the implanted gestational sac and protrudes into the endometrial lumen It represents the maternal decidual reaction and the beginning of maternal-fetal circulation. This area is also believed to be responsible for future placental formation and development (Brosens and Gellersen, 2010) Distance between the implantation site and the internal cervical ostium (os). This was taken from the lower end of the hyperechoic trophoblast ring of the gestational sac to the internal cervical os in the sagittal plane.

         * doppler assessment of the retro chorionic blood flow in the area behind the maximum chorionic tissue to detect sensitivity index (RI),in cases of low gestational sac Doppler assessment of peri trophoplastic blood flow will be assessed.
   2. then the patient will be enrolled during routine ANC till delivery and data collected at32-34 weeks gestation regarding placental site will be correlated with 1st data and data at delivery

DETAILED DESCRIPTION:
After gaining verbal consent , Patients included in this study will be subjected to:

1. history taking :

   * peronal history .
   * obstetric history.
   * past history
2. general examination including vital signs
3. abominal and pelvic examination
4. the patient will be examined son graphically at 3 visits

   1. The first visit at less than 10 weeks gestation :trans vaginal ultrasound with partially filled bladder to nullify effect of anteversion of the uterus for assessment of---the site of the intrauterine gestational sac in relation to the endometrial cavity . For the purposes of this study and to obtain consistent findings, it was decided to have only five subgroups of gestational site implantation in relation to the endometrial cavity (Fig. 2):

      1. anterior,
      2. posterior,
      3. Fundal,
      4. low-lying anterior,\
      5. low lying posterior

      We adopted the definition of implantation site from previous publication (Abdallah et al., 2012). The implantation site is visualized in the sagittal plane as a hyperechoic ring that occupies one side of the implanted gestational sac and protrudes into the endometrial lumen It represents the maternal decidual reaction and the beginning of maternal-fetal circulation. This area is also believed to be responsible for future placental formation and development (Brosens and Gellersen, 2010) Distance between the implantation site and the internal cervical ostium (os). This was taken from the lower end of the hyperechoic trophoblast ring of the gestational sac to the internal cervical os in the sagittal plane.

      -----doppler assessment of the retro chorionic blood flow in the area behind the maximum chorionic tissue to detect sensitivity index (RI),in cases of low gestational sac Doppler assessment of peri trophoplastic blood flow will be assessed.
   2. then the patient will be enrolled during routine ANC till delivery and data collected at32-34 weeks gestation regarding placental site will be correlated with 1st data and data at delivery

ELIGIBILITY:
Inclusion Criteria:

* singleton intrauterine pregnancy.
* gestational age less than 10 weeks
* history of previous cesarean section(one or more)

Exclusion Criteria:

* negative fetal pole pulsation.
* any condition distorting uterine cavity i.e uterine myoma,uterine cavity anomalies
* multifetal pregnancy.
* any condition necessitate termination of early pregnancy i.e maternal medical disorder ,molar pregnancy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: pregnant women with or without previous cesarean section scar are assessed at 10 weeks of gestational age then at 36 weeks to detect the relation between implantation site and placental site
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-15 (Estimated); Primary Completion 2018-08-31 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Placenta previa | at 36 weeks of gestational age
  measuring the distance between lower placental edge and internal os of the cervix by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, MD, Principal Investigator — kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided